CLINICAL TRIAL: NCT03012022
Title: Nitrative Stress in Heart Failure: The Cleveland Heart and Metabolic Prevention Study (CHAMPS)
Brief Title: Cleveland Heart and Metabolic Prevention Study
Acronym: CHAMPS
Status: Active, not recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Wilson Tang, Principal Investigator, Staff Cellular and Molecular Medicine and Cardiovascular Medicine, The Cleveland Clinic, The Cleveland Clinic
Other Study IDs: 10-727; 1R01HL103931 (NIH)
Record Dates: First submitted 2016-12-15; First posted 2017-01-06 (Estimated); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Heart Failure Risk Factors in Healthy Individuals
Keywords: Healthy Volunteers; Congestive Heart Failure; Cardiomyopathies; Heart Failure; Risk Factors
MeSH Terms: conditions — Heart Failure; Cardiomyopathies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood, Serum, Plasma, Red Blood Cells, Buffy Coat, Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Volunteers: Volunteers without known cardiomyopathy or heart failure

SUMMARY:
The purpose of this research study is to investigate the role of chemical reactions, such as inflammation and oxidation, in the cause of cardiac dysfunction (the heart does not function properly). The investigators are interested in studying the various chemical pathways for cell damage to determine which are the most prevalent and/or most important. The investigators also want to determine whether waste products of oxidative damage or other chemicals can be monitored in the blood or urine and serve as an indication of the existence and severity of overall heart disease activity. The investigators further want to determine whether certain proteins, called enzymes, affect this cell damage, or whether the presence or absence of certain genes which create different forms of these enzymes correlate with the development of heart failure or cardiomyopathy (weakening of the heart muscle or a change in heart muscle structure) or other cardiovascular diseases.

DETAILED DESCRIPTION:
This is a single-center study conducted at the Cleveland Clinic. The target population for this study is very broad and goes beyond any specific cohort or community. Participants will be mainly recruited from the greater Cleveland/Akron area, but any volunteer meeting the inclusion/exclusion criteria is eligible for participation.

The overall goal of the Cleveland Heart And Metabolic Prevention Study (CHAMPS) is to determine the role of nitrative stress in the development and progression of heart failure (HF) and left ventricular systolic dysfunction (LVSD). The investigators have previously developed and performed preliminary clinical validation studies on multiple specific molecular footprints of known pathways of nitric oxide (NO) pathobiology that affect substrate availability for NO production or generation of NO-derived oxidants as a result of nitrative stress. For each these molecular markers and indices, mechanistic links to cardiovascular diseases have been demonstrated. However, these processes may be differentially expressed in different proportions at different stages of LVSD/HF disease progression, and certainly may vary among different individuals. It is the investigators' hypothesis that the interplay of many of these processes contribute to development of subclinical myocardial dysfunction (SMD), and the progression to overt LVSD and HF.

In order to help determine the role of nitrative stress in the development and progression of heart failure and left ventricular systolic dysfunction study participants will receive many non-invasive, research only, procedures as well as a blood draw and urine collection. The procedures performed may include electrocardiogram (ECG), echocardiogram, carotid intima-medial thickness measurements, ankle-brachial index, bioelectrical impedance analysis, pulse wave velocity analysis, spirometry, exhaled nitric oxide analysis, and venous occlusion strain-gauge plethysmography. The specific tests performed on each participant will be at the description of the primary investigator and not all participants will receive all tests. All participants will have blood and urine collections and all participants will be asked to fill out questionnaires pertaining to family history, personal medical history and estimates of functional capacity.

Specific aims include:

Aim 1: To test the hypothesis that levels of specific nitric oxide (NO)-mediated processes are associated with the presence of SMD and LVSD/HF.

Aim 2: To test the hypothesis that levels of specific NO-mediated processes are associated with prospective risks for development of adverse cardiovascular events and overt HF in stable patients without LVSD/HF at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Either age 40 years or older OR age 18 years or older with a family history of heart failure or cardiac dysfunction (the heart does not function properly).
* Able and willing to consent to the study protocol, including an overnight (≥10 hour) fast.

Exclusion Criteria:

* Known history of heart failure or cardiomyopathy (LVSD, defined by left ventricular ejection fraction ≤45%) at the time of enrollment
* Major cardiovascular event (myocardial infarction, unstable angina, stroke, transient ischemic attack, pulmonary embolism), or major surgery <1 month of enrollment of present study (subject can be considered enrollment after 1 month if deemed clinically stable)
* Any hospitalization or emergency room visits for any cause <1 month of enrollment present study
* Known life expectancy <6 months at the time of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 1208 (Actual)
Dates: Start 2010-11-08 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Correlation between metabolic and/or nitrative stress markers and predefined clinical endpoints | 10 years
  Clinical endpoints include acute myocardial infarction, acute coronary syndrome, congestive heart failure, serious cardiac arrhythmia, peripheral vascular disease, cerebrovascular events and death. Events will be aggregated into a common category (e.g. MACE) for statistical analysis and reporting. These aggregated events data will then be correlated with each biomarker of interest.

SECONDARY OUTCOMES:
Determination of sub-clinical myocardial dysfunction by echocardiogram | 10 years
  Determination of sub-clinical myocardial dysfunction by echocardiogram
Correlation between DASI functional capacity and markers of metabolic and nitrative stress | 10 years
  Correlation between functional capacity, as measured by the Duke Activity Status Index (DASI) questionnaire, and markers of metabolic and nitrative stress
Correlation between SF36 functional capacity and markers of metabolic and nitrative stress | 10 years
  Correlation between functional capacity, as measured by the SF36 version 2 questionnaire, and markers of metabolic and nitrative stress
Correlation between DASI functional capacity and markers of cardiac dysfunction | 10 years
  Correlation between functional capacity, as measured by DASI questionnaire, and markers of cardiac dysfunction
Correlation between SF36 functional capacity and markers of cardiac dysfunction | 10 years
  Correlation between functional capacity, as measured by SF36 version 2 questionnaire, and markers of cardiac dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: W. H. Wilson Tang, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abu-Soud HM, Hazen SL. Nitric oxide is a physiological substrate for mammalian peroxidases. J Biol Chem. 2000 Dec 1;275(48):37524-32. doi: 10.1074/jbc.275.48.37524. PMID 11090610
- [Background] Shiva S, Wang X, Ringwood LA, Xu X, Yuditskaya S, Annavajjhala V, Miyajima H, Hogg N, Harris ZL, Gladwin MT. Ceruloplasmin is a NO oxidase and nitrite synthase that determines endocrine NO homeostasis. Nat Chem Biol. 2006 Sep;2(9):486-93. doi: 10.1038/nchembio813. Epub 2006 Aug 13. PMID 16906150
- [Background] Tang WH, Wang Z, Cho L, Brennan DM, Hazen SL. Diminished global arginine bioavailability and increased arginine catabolism as metabolic profile of increased cardiovascular risk. J Am Coll Cardiol. 2009 Jun 2;53(22):2061-7. doi: 10.1016/j.jacc.2009.02.036. PMID 19477356
- [Background] Mullens W, Abrahams Z, Francis GS, Sokos G, Starling RC, Young JB, Taylor DO, Tang WH. Usefulness of Isosorbide Dinitrate and Hydralazine as add-on therapy in patients discharged for advanced decompensated heart failure. Am J Cardiol. 2009 Apr 15;103(8):1113-9. doi: 10.1016/j.amjcard.2008.12.028. Epub 2009 Feb 21. PMID 19361599
- [Background] Taylor AL, Ziesche S, Yancy C, Carson P, D'Agostino R Jr, Ferdinand K, Taylor M, Adams K, Sabolinski M, Worcel M, Cohn JN; African-American Heart Failure Trial Investigators. Combination of isosorbide dinitrate and hydralazine in blacks with heart failure. N Engl J Med. 2004 Nov 11;351(20):2049-57. doi: 10.1056/NEJMoa042934. Epub 2004 Nov 8. PMID 15533851
- [Background] Hare JM, Colucci WS. Role of nitric oxide in the regulation of myocardial function. Prog Cardiovasc Dis. 1995 Sep-Oct;38(2):155-66. doi: 10.1016/s0033-0620(05)80004-0. PMID 7568904
- [Background] Elahi MM, Naseem KM, Matata BM. Nitric oxide in blood. The nitrosative-oxidative disequilibrium hypothesis on the pathogenesis of cardiovascular disease. FEBS J. 2007 Feb;274(4):906-23. doi: 10.1111/j.1742-4658.2007.05660.x. Epub 2007 Jan 22. PMID 17244198
- [Background] Champion HC, Skaf MW, Hare JM. Role of nitric oxide in the pathophysiology of heart failure. Heart Fail Rev. 2003 Jan;8(1):35-46. doi: 10.1023/a:1022142904202. PMID 12652158
- [Background] Recchia FA. Role of nitric oxide in the regulation of substrate metabolism in heart failure. Heart Fail Rev. 2002 Apr;7(2):141-8. doi: 10.1023/a:1015324508556. PMID 11988638
- [Background] Mullens W, Abrahams Z, Francis GS, Skouri HN, Starling RC, Young JB, Taylor DO, Tang WH. Sodium nitroprusside for advanced low-output heart failure. J Am Coll Cardiol. 2008 Jul 15;52(3):200-7. doi: 10.1016/j.jacc.2008.02.083. PMID 18617068
- [Background] Carson P, Ziesche S, Johnson G, Cohn JN. Racial differences in response to therapy for heart failure: analysis of the vasodilator-heart failure trials. Vasodilator-Heart Failure Trial Study Group. J Card Fail. 1999 Sep;5(3):178-87. doi: 10.1016/s1071-9164(99)90001-5. PMID 10496190
- [Background] Vanderheyden M, Bartunek J, Knaapen M, Kockx M, De Bruyne B, Goethals M. Hemodynamic effects of inducible nitric oxide synthase and nitrotyrosine generation in heart failure. J Heart Lung Transplant. 2004 Jun;23(6):723-8. doi: 10.1016/j.healun.2003.07.015. PMID 15366433
- [Background] Pacher P, Schulz R, Liaudet L, Szabo C. Nitrosative stress and pharmacological modulation of heart failure. Trends Pharmacol Sci. 2005 Jun;26(6):302-10. doi: 10.1016/j.tips.2005.04.003. PMID 15925705
- [Background] Reinartz M, Ding Z, Flogel U, Godecke A, Schrader J. Nitrosative stress leads to protein glutathiolation, increased s-nitrosation, and up-regulation of peroxiredoxins in the heart. J Biol Chem. 2008 Jun 20;283(25):17440-9. doi: 10.1074/jbc.M800126200. Epub 2008 Apr 21. PMID 18426799
- [Background] Ungvari Z, Gupte SA, Recchia FA, Batkai S, Pacher P. Role of oxidative-nitrosative stress and downstream pathways in various forms of cardiomyopathy and heart failure. Curr Vasc Pharmacol. 2005 Jul;3(3):221-9. doi: 10.2174/1570161054368607. PMID 16026319
- [Background] Shishehbor MH, Aviles RJ, Brennan ML, Fu X, Goormastic M, Pearce GL, Gokce N, Keaney JF Jr, Penn MS, Sprecher DL, Vita JA, Hazen SL. Association of nitrotyrosine levels with cardiovascular disease and modulation by statin therapy. JAMA. 2003 Apr 2;289(13):1675-80. doi: 10.1001/jama.289.13.1675. PMID 12672736
- [Background] Shishehbor MH, Brennan ML, Aviles RJ, Fu X, Penn MS, Sprecher DL, Hazen SL. Statins promote potent systemic antioxidant effects through specific inflammatory pathways. Circulation. 2003 Jul 29;108(4):426-31. doi: 10.1161/01.CIR.0000080895.05158.8B. Epub 2003 Jul 14. PMID 12860913
- [Background] Hazen SL, Zhang R, Shen Z, Wu W, Podrez EA, MacPherson JC, Schmitt D, Mitra SN, Mukhopadhyay C, Chen Y, Cohen PA, Hoff HF, Abu-Soud HM. Formation of nitric oxide-derived oxidants by myeloperoxidase in monocytes: pathways for monocyte-mediated protein nitration and lipid peroxidation In vivo. Circ Res. 1999 Nov 12;85(10):950-8. doi: 10.1161/01.res.85.10.950. PMID 10559142
- [Background] Abu-Soud HM, Hazen SL. Nitric oxide modulates the catalytic activity of myeloperoxidase. J Biol Chem. 2000 Feb 25;275(8):5425-30. doi: 10.1074/jbc.275.8.5425. PMID 10681518
- [Background] Podrez EA, Schmitt D, Hoff HF, Hazen SL. Myeloperoxidase-generated reactive nitrogen species convert LDL into an atherogenic form in vitro. J Clin Invest. 1999 Jun;103(11):1547-60. doi: 10.1172/JCI5549. PMID 10359564
- [Background] Parastatidis I, Thomson L, Fries DM, Moore RE, Tohyama J, Fu X, Hazen SL, Heijnen HF, Dennehy MK, Liebler DC, Rader DJ, Ischiropoulos H. Increased protein nitration burden in the atherosclerotic lesions and plasma of apolipoprotein A-I deficient mice. Circ Res. 2007 Aug 17;101(4):368-76. doi: 10.1161/CIRCRESAHA.107.157537. Epub 2007 Jul 5. PMID 17615369
- [Background] Leeuwenburgh C, Hardy MM, Hazen SL, Wagner P, Oh-ishi S, Steinbrecher UP, Heinecke JW. Reactive nitrogen intermediates promote low density lipoprotein oxidation in human atherosclerotic intima. J Biol Chem. 1997 Jan 17;272(3):1433-6. doi: 10.1074/jbc.272.3.1433. PMID 8999808
- [Background] Zheng L, Nukuna B, Brennan ML, Sun M, Goormastic M, Settle M, Schmitt D, Fu X, Thomson L, Fox PL, Ischiropoulos H, Smith JD, Kinter M, Hazen SL. Apolipoprotein A-I is a selective target for myeloperoxidase-catalyzed oxidation and functional impairment in subjects with cardiovascular disease. J Clin Invest. 2004 Aug;114(4):529-41. doi: 10.1172/JCI21109. PMID 15314690
- [Background] Wu Z, Wagner MA, Zheng L, Parks JS, Shy JM 3rd, Smith JD, Gogonea V, Hazen SL. The refined structure of nascent HDL reveals a key functional domain for particle maturation and dysfunction. Nat Struct Mol Biol. 2007 Sep;14(9):861-8. doi: 10.1038/nsmb1284. Epub 2007 Aug 5. PMID 17676061
- [Background] Brennan ML, Penn MS, Van Lente F, Nambi V, Shishehbor MH, Aviles RJ, Goormastic M, Pepoy ML, McErlean ES, Topol EJ, Nissen SE, Hazen SL. Prognostic value of myeloperoxidase in patients with chest pain. N Engl J Med. 2003 Oct 23;349(17):1595-604. doi: 10.1056/NEJMoa035003. PMID 14573731
- [Background] Vita JA, Brennan ML, Gokce N, Mann SA, Goormastic M, Shishehbor MH, Penn MS, Keaney JF Jr, Hazen SL. Serum myeloperoxidase levels independently predict endothelial dysfunction in humans. Circulation. 2004 Aug 31;110(9):1134-9. doi: 10.1161/01.CIR.0000140262.20831.8F. Epub 2004 Aug 23. PMID 15326065
- [Background] Meuwese MC, Stroes ES, Hazen SL, van Miert JN, Kuivenhoven JA, Schaub RG, Wareham NJ, Luben R, Kastelein JJ, Khaw KT, Boekholdt SM. Serum myeloperoxidase levels are associated with the future risk of coronary artery disease in apparently healthy individuals: the EPIC-Norfolk Prospective Population Study. J Am Coll Cardiol. 2007 Jul 10;50(2):159-65. doi: 10.1016/j.jacc.2007.03.033. Epub 2007 Jun 21. PMID 17616301
- [Background] Tang WH, Tong W, Shrestha K, Wang Z, Levison BS, Delfraino B, Hu B, Troughton RW, Klein AL, Hazen SL. Differential effects of arginine methylation on diastolic dysfunction and disease progression in patients with chronic systolic heart failure. Eur Heart J. 2008 Oct;29(20):2506-13. doi: 10.1093/eurheartj/ehn360. Epub 2008 Aug 6. PMID 18687662